CLINICAL TRIAL: NCT05390177
Title: Memory for Health Research Findings
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never started because it was not funded; the study will not be conducted unless funded in the future
Sponsor: University of Colorado, Colorado Springs (Other)
Responsible Party: Principal Investigator, Lori James, Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 22-011
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Healthy Aging

STUDY DESIGN:
Intervention Model Description: Participants from two age groups (young vs. older adults) will be compared for two experimental conditions. Although age group cannot be randomly assigned, the comparison between groups makes the design factorial.
Who Masked: Participant
Masking Description: Participants are unaware which study condition they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First health video (Experimental): This video presents health information for one study condition.
  Interventions: Behavioral: Video type
- Second health video (Active Comparator): This video presents health information for one study condition.
  Interventions: Behavioral: Video type

INTERVENTIONS:
Behavioral: Video type — One of two videos presenting health research findings (each 2.5 minutes in length) will be shown to a participant.

SUMMARY:
This experiment tests young (ages 18-35) and older adult (ages 60-80) participants. Participants will watch a brief video, will complete a memory task, and will complete measures about their beliefs.

DETAILED DESCRIPTION:
Participants (360 young adults and 360 older adults) will complete a baseline beliefs measure and will then be randomly assigned to one of two study conditions. They will watch a 2.5-min video that presents research findings related to their health. Their memory for the video will be tested, and participants will also complete a demographic questionnaire and another survey about their beliefs. Participation will last 15-20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years old or 60 to 80 years old
* Fluent English speakers

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Health Beliefs | 3 minutes
  A survey about the participant's beliefs

CONTACTS AND LOCATIONS:
Overall Officials: Lori James, PhD, Principal Investigator — University of Colorado, Colorado Springs
Locations (1):
- UCCS, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from individual participants will be shared (e.g., via OSF) if required for publication or requested by other researchers.
Time Frame: It will be shared at the time of publication and available indefinitely
Access Criteria: De-identified data will be publicly available if required for publication.